CLINICAL TRIAL: NCT00390091
Title: A Randomized, Double-Blind Study to Evaluate the Safety, Pharmacokinetic and Pharmacodynamic Effects of Abetimus Sodium in Patients With Systemic Lupus Erythematosus (SLE)
Brief Title: Study of LJP 394 (Abetimus Sodium) in Lupus Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: La Jolla Pharmaceutical Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: LJP 394-90-16
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2007-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; Nephritis; Kidney; SLE; Systemic Lupus Erythematosus; Nephritis, Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Nephritis; Lupus Nephritis | interventions — abetimus

INTERVENTIONS:
Drug: abetimus sodium (LJP 394)

SUMMARY:
The primary purpose of this study is to assess the safety and pharmacodynamic effect of LJP 394 at doses of 100 mg, 300 mg and 900 mg on anti-dsDNA antibody levels in patients with SLE.

DETAILED DESCRIPTION:
STUDY NOW INCORPORATED INTO PHASE 3 STUDY NCT00089804.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 12 and 70 years old.
* Diagnosis of Systemic Lupus Erythematosus (SLE)
* Females must be non-pregnant and non-lactating. Females must agree to use adequate birth control methods during the course of the study.
* Ability to have weekly intravenous (IV) administration of study drug.

Exclusion Criteria:

* Prior exposure to abetimus sodium within 6 months prior to screening.
* Patients not on stable medications for 30 days prior to screening.
* Patients with acute or chronic infections.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-09

PRIMARY OUTCOMES:
The assessment of the safety and pharmacodynamic effect of abetimus sodium at
doses of 100mg, 300mg, and 900mg in reducing the anti-dsDNA antibody levels in
patients with SLE will be based on laboratory data from the central laboratory
and confirmed by supporting data. The pharmacodynamic effic will be assessed
using historical placebo effect as a control.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Linnik, PhD, Study Chair — La Jolla Pharmaceutical Company
Locations (2):
- United States (2):
  - Wallace Rheumatic Study Center, Los Angeles, California
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania

REFERENCES:
- See also: Sponsor's website — http://www.ljpc.com
- See also: STUDY NOW INCORPORATED INTO PHASE 3 STUDY NCT00089804 — http://clinicaltrials.gov/ct/show/NCT00089804?order=1